CLINICAL TRIAL: NCT04945525
Title: A Patient Self-Assessment Software Combining Compliance Protocols to Improve Prescriber Confidence, Reduce Liability, and Improve Patient Outcomes
Brief Title: Comparing a Patient Self-Assessment Software to Treatment as Usual in Opioid Prescriber and Patient Opioid Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sure Med Compliance (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1289337; 1R44DA051272-01 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Opioid-use Disorder; Opioid Misuse; Opioid Use; Chronic Pain
Keywords: Pain; Pain Management; Patient Risk; Patient-Focused Outcomes; Outcomes Research; Patient Care; Self Assessment; Digital; Opioid Epidemic; Opioid Misuse; Patient Safety; Prescription Opioid; Software Development; Opioid Prescriber; Documentation; Legitimate Medical Purpose; Computer Software; Electronic Health Record; Laws; Monitor; Medication Compliance; Intervention; Chart Documentation; Prescriber Confidence; NIH Heal Initiative
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain; Pain; Agnosia; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Forty-six clinics with chronic, non-cancer pain patients in both pain management and general practice settings will be randomized to the Care Continuity Program (CCP) intervention or control group. Both groups will view an Accreditation Council for Continuing Medical Education (ACCME) accredited educational video about the safe initiation, continuation, and discontinuation of opioid therapy, as well as the data elements required by law and regulation to be included in the medical records of patients prescribed opioids. After four months of intervention, the CCP's ability to lower morphine milligram equivalents (MME), improve physical functioning in patients, mitigate the opioid prescriber's legal risk, and increase confidence levels in opioid prescribing among prescribers will be measured by completing medical record audits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care Continuity Program + Education (Experimental): Participating clinics (and their prescribers and patients) will be randomly selected to implement the Care Continuity Program (CCP) intervention, at which time prescribers will view an Accreditation Council for Continuing Medical Education (ACCME) accredited educational video about the safe initiation, continuation, and discontinuation of opioid therapy, as well as the data elements required by law and regulation to be included in the medical records of patients prescribed opioids. Then patients will receive welcome letters and be required to complete CCP self-assessments before each appointment. Prescribers will begin using the generated CCP summary page at each appointment to help make decisions about initiating or maintaining an opioid prescription for an individual patient.
  Interventions: Other: Care Continuity Program
- Education Alone (No Intervention): Participating clinics (and their prescribers and patients) will be randomly selected to the control group, at which time prescribers will view an Accreditation Council for Continuing Medical Education (ACCME) accredited educational video about the safe initiation, continuation, and discontinuation of opioid therapy, as well as the data elements required by law and regulation to be included in the medical records of patients prescribed opioids. Then patients and prescribers will continue treatment as usual in their clinic.

INTERVENTIONS:
Other: Care Continuity Program — The Care Continuity Program is an online patient self-assessment tool used by prescribers of opioids to better identify patient risk factors and opioid therapy benefit. This tool is completed by the patient, outside of the office, using an internet enabled device and follows a compliance driven protocol developed by analyzing case law against physicians in mis-prescribing opioid cases. Results, in the form of a date and time stamped legal report, are instantly transmitted to the prescriber's electronic health records, mitigating the prescriber's civil and criminal risk. A brief of findings is displayed within the software through a dashboard and on the summary page of the report. Prescribers may use the summary page to help them identify the appropriateness of initiating opioid therapy and/or continuing opioid therapy.
  Arms: Care Continuity Program + Education

SUMMARY:
The Care Continuity Program (CCP), a product of Sure Med Compliance, is a novel, online patient self-assessment used by prescribers of opioids to better identify patient risk factors and therapy benefit. This tool is completed by the patient, outside of the office, using an internet enabled device and follows a compliance driven protocol developed by analyzing case law against physicians in mis-prescribing opioid cases. Results, in the form of a date and time stamped legal report, are instantly transmitted to the prescriber's electronic health records, mitigating the prescriber's civil and criminal risk. A brief of findings is displayed within the software through a dashboard and on the summary page of the report. This software offering includes a mobile and standard web-based application. The objective of the proposed research is to validate the protocols and delivery system of the CCP by measuring patient outcomes, prescriber confidence, and completeness of documentation in the patient chart in primary care and pain management settings, pre and post implementation of the CCP.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed an opioid at a participating clinic
* Completed a baseline CCP assessment
* Report functional impairment due to chronic pain
* Report at least a 4 out of 10 on pain intensity
* Have no psychiatric, mental, or physical limitation that precludes participation in the trial

Exclusion Criteria:

* Current cancer diagnosis
* Palliative or end of life care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1840 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Morphine Milligram Equivalent | Approximately 4 Months
  This is a measure of the dosage of opioid medication prescribed, with higher Morphine Milligram Equivalent (MME) representing higher dosage. For this project, MME will be calculated using the Centers for Disease Control and Prevention Opioid Guidelines smartphone app, which includes an MME calculator. We will compare average MME of the groups at the end of the four month intervention.
Physical Functioning | Approximately 4 Months
  In a survey adapted from the PDI (pain disability index) and the BPI (brief pain inventory) interference items, patients rate how much difficulty they have had in the past two weeks with each of seven life activity categories (family/home responsibilities, recreational activities, social activities, work-related activities, sex life, self-care activities, and life-supporting activities) because of pain. These items are measured from 0-10.
Prescriber Risk | Approximately 4 Months
  Prescriber risk will be assessed as the completion of 26 data elements including: pain measurement, physical functional impairment, physical exam, onset of pain, duration of pain, failure on alternate treatment, assessment of affect, PTSD screening, assessment of substance use disorder risk, assessment of alcohol use, drug testing, consulting of state prescription drug monitoring program, patient history, informed consent to opioid therapy, controlled substance agreement, patient opioid education, treatment goals properly established, opioids initiated properly, starting MME under 90, no concomitant benzodiazepine use, side effects or adverse events evaluation, patient seen in office with proper frequency based on risk, opioid use disorder patients referred for treatment, and patient stratified into level of risk for misuse. At the end of the 4 month intervention, we will compare the proportion of each group's medical encounter notes that are complete.
Prescriber Confidence | Approximately 4 Months
  This outcome will be assessed via a survey developed based on the Opioid Therapy Survey (OTS). Our survey is a 19-item questionnaire that assesses prescriber confidence and fear of regulatory, civil, and criminal investigations. The post-intervention survey includes an additional 5 items on the effectiveness of the Care Continuity Program. At the end of the 4 month intervention, we will compare average prescriber confidence scores between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Hartzema, PhD, Principal Investigator — Sure Med Compliance; John Bowman, BS, Study Director — Sure Med Compliance
Locations (1):
- Sure Med Compliance, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
As an NIH Helping to End Addiction Long-Term (HEAL) Initiative study, we are committed to making our publications and data available to researchers. Electronic copies of publications will be deposited (within four weeks of acceptance by a journal) in PubMed Central with proper metadata to be made discoverable and accessible upon publication. Publications will be made publicly available immediately without any embargo period. Underlying primary data for the publications that are free of identifiers but contain sensitive information will be made broadly available through the NIH HEAL Initiative central data repository. Underlying primary data will be deposited in the NIH HEAL Initiative central data repository after it is stripped of all identifiers in accordance with HIPAA regulations and the Department of Health and Human Services Regulations for the Protection of Human Subjects to ensure that the identities of research subjects cannot be readily ascertained from the data.